CLINICAL TRIAL: NCT02314208
Title: Therapeutic Metabolic Intervention in Patients With Spastic Paraplegia SPG5
Acronym: SPA-M
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C14-04
Record Dates: First submitted 2014-11-14; First posted 2014-12-11 (Estimated); Last update posted 2025-09-02 (Actual); Status verified 2025-02

CONDITIONS: Spastic Paraplegia, Hereditary
Keywords: spastic paraplegia; metabolism; oxysterols; neurogenetics
MeSH Terms: conditions — Spastic Paraplegia, Hereditary; Paraplegia | interventions — Chenodeoxycholic Acid; Resveratrol; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Xenbilox (Active Comparator): Xenbilox (chenodeoxycholic acid) 1000mg capsule by mouth every day for 2 months
  Interventions: Drug: Xenbilox
- Resveratrol (Active Comparator): Resveratrol 80mg capsule by mouth every day for 2 months
  Interventions: Dietary Supplement: Resveratrol
- Tahor (Active Comparator): Tahor (atorvastatin) 40mg tablet by mouth every day for 2 months
  Interventions: Drug: Tahor

INTERVENTIONS:
Drug: Xenbilox
  Other Names: Chenodeoxycholic acid
  Arms: Xenbilox
Dietary Supplement: Resveratrol
  Arms: Resveratrol
Drug: Tahor
  Other Names: Atorvastatin
  Arms: Tahor

SUMMARY:
The purpose of this project is to study the efficacy of three candidate molecules (Xenbilox, Tahor and Resveratrol) in order to decrease the production of oxysterols by reducing the synthesis of cholesterol and/or regulate the production of bile acids and/or enabling neuroprotective action within the motor neuron.

DETAILED DESCRIPTION:
The primary objective of the study is:

- decrease the accumulation of metabolites which can have a negative impact on neurological and systemic function of patients with SPG5.

The secondary objectives of the study are:

* confirm the clinical and biological tolerance of the different candidate molecules under study
* improve the serum bile acid profile of patients with SPG5

ELIGIBILITY:
Inclusion Criteria:

* patients that have confirmed through genetic testing their status as carriers of 2 mutations in the CYP7B1 gene
* age ≥ 18 years
* patients that have signed the informed consent form
* presence of health care coverage

Exclusion Criteria:

* known hypersensitvity to chenodeoxycholic acid, atorvastatin, resveratrol or to any of their byproducts
* cholesterol lowering medications other than the study treatment
* hepatic failure with transaminases >3 times the normal level
* progressive biliary pathology
* chronic diarrhea
* serious mental illness
* significant comorbid neurological disorder
* incapacity to understand information about the protocol
* unwilling or unable to participate in any part of the study
* participation in another clinical trial during the study period
* person deprived of liberty by judicial or administrative decision
* adult subject under legal protection or unable to consent
* pregnant or breastfeeding women
* lack of health care coverage
* absence of a signed informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-01-08 (Actual); Primary Completion 2017-09-27 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Change of 27-hydroxycholesterol blood level after 2 months of treatment for each treatment | 2 months
  27-hydroxycholesterol will be measured on fasten blood samples for the 12 patients included before and after the 2-month treatment period for each treatment

SECONDARY OUTCOMES:
Modification of the serum acid profile after a 2-month treatment measured in blood and urine samples | 2 months
  In blood and urines samples of the 12 patients, the following criteria will be assesed in order to observe an evolution of the acid profile:
  * total biliary acids
  * ratio of primary/secondary biliary acids
  * the ratio cholic acids/chenodeoxycholic acids
  * the ratio chenodeoxycholic acids/ lithocholic acids
Change of 25-hydroxycholesterol blood level after 2 months of treatment for each treatment | 2 months
  25-hydroxycholesterol will be measured on fasten blood samples for the 12 patients included before and after the 2-month treatment period for each treatment
Number of participants with adverse events related with digestive problems | 18 months
  During the study, adverse events related with digestive problems will be evaluate in order to asses the clinical tolerance to each treatment
Number of partcipants with adverse events related with standard biological parameters | 18 months
  Biological tolerance will be evaluate on patients blood samples at each visit. The following criteria will be assessed:
  * ionogram and fasting glucose
  * kidney and liver function with urea, creatinine,lipase, amylase, bilirubine, creatine phosphokinase, transaminases,sodium, potassium, calcium, phosphorus

CONTACTS AND LOCATIONS:
Overall Officials: Fanny MOCHEL, MD-PhD, Principal Investigator — Pitié-Salpêtrière Hospital
Locations (1):
- Pitié-Salpêtrière Hospital, Paris, France

REFERENCES:
- [Background] Marelli C, Lamari F, Rainteau D, Lafourcade A, Banneau G, Humbert L, Monin ML, Petit E, Debs R, Castelnovo G, Ollagnon E, Lavie J, Pilliod J, Coupry I, Babin PJ, Guissart C, Benyounes I, Ullmann U, Lesca G, Thauvin-Robinet C, Labauge P, Odent S, Ewenczyk C, Wolf C, Stevanin G, Hajage D, Durr A, Goizet C, Mochel F. Plasma oxysterols: biomarkers for diagnosis and treatment in spastic paraplegia type 5. Brain. 2018 Jan 1;141(1):72-84. doi: 10.1093/brain/awx297. PMID 29228183